CLINICAL TRIAL: NCT05812144
Title: New Clinical Outcome Measures to Remotely Evaluate Patients With FacioScapuloHumeral Muscular Dystrophy - PROGRESS FSHD
Brief Title: New Clinical Outcome Measures to Remotely Evaluate Patients With FacioScapuloHumeral Muscular Dystrophy
Acronym: PROGRESS-FSHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-PP-01
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Facioscapulohumeral Muscular Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with type 1 facioscapulohumeral muscular dystrophy (Other)
  Interventions: Other: Remote monitoring program

INTERVENTIONS:
Other: Remote monitoring program — Remote program is composed of some questionnaires and physical exercises performed at home and at hospital (depending on the concerned visit)

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSHD) is one of the most common adult muscular dystrophy with an estimated prevalence range of 2-7 per 100,000. The disease is characterized by slowly progressive, asymmetric muscle weakness that starts with the face and scapular muscles. It causes significant lifetime morbidity, with up to 20% of patients eventually requiring full-time wheelchair use. However, there is a large degree of clinical variability in both disease progression and severity. This makes predicting an individual's disease course difficult and has made clinical trial design and the development of new therapeutic strategies challenging.

The disease is caused by the aberrant expression of a normally silenced gene, Double homeobox 4 (DUX4), which causes disease by a toxic gain-of-function. The emergence of the pathophysiologic model provided several possible therapeutic approaches to treat FSHD. However, as drugs move from preclinical testing into human trials, it is essential to validate clinical trial tools and methodologies to facilitate drug development from early phase studies through registration trials. Natural history studies are conducted to develop and validate new clinical outcome measures (COMs). A large international multicenter study is currently ongoing in order to validate COMs in ambulant FSHD patients (ReSolve, NCT03458832). Additionally, Nice University Hospital is conducting an ancillary study (CTRN FSHD France, NCT04038138) to evaluate muscle MRI, an additional emerging biomarker, to follow disease progression in the same patient population.

Nevertheless, these studies are focused on the development of COMs collected at the hospital. In this setting, several factors that may interfere with disease progression or patient quality of life are underestimated (daily exercise, daily pain or fatigue, the psychological impact of the disease, and falls…). Consequently, and given the context of the current pandemic, the interest of pharmaceutical companies, stakeholders, clinicians, and researchers in data collected in a cohort of FSHD patients at home is rapidly increasing. Consequently, a new battery of COMs adapted for the remote evaluation needs to be developed and/or validated. There are clear benefits to remote assessments. The ability to observe an individual perform functional mobility tasks and self-care in their natural environment is meaningful and invaluable.

The set-up of a reliable remote assessment will allow for ensuring drug home delivery, maintaining patients on trials, and collecting and analysing additional data to improve patient stratification in clinical trials and develop new approaches to assess the short-term and long-term efficacy of a given therapy. Remote assessment can also be the key to developing more efficient real-life studies, empowering patients and caregivers in the management of this disease, and more efficiently monitoring drug side effects or the socio-economic burden of the disease. The overall aim of the PROGRESS FSHD study is to experiment the feasibility of the remote evaluation in patients with FSHD, through the use of a patient-oriented mobile application (myFSHD app). The content of the application has been determined after extensive discussions with patients and patients' associations that have identified their unmet needs and based on preliminary results of the CTRN FSHD France project. The video-recorded exercises have been designed specifically to stress a particular body region. The myFSHD mobile application will be used by 70 FSHD1 patient during 12 months, at home and at the hospital, to administer patient-reported questionnaires on fatigue, pain, physical activity, sleep, quality of life, and socio-economic burden of the disease, as well as video of validated scores and scales. The collected data will help to:

* Evaluate patients' adherence to the program
* Evaluate the technical feasibility of remote evaluation
* Assess the reliability of remote evaluation
* Assess the robustness of new COMs compared to commonly used COMs
* Evaluate the quality of life and socio-economic burden of the disease Overall, this study will provide digital tools adapted to monitor disease evolution remotely in FSHD patients. The patient-generated measures collected through connected digital tools (patient full-body motion videos collected through the myFSHD app) can be used to explain, influence, and/or predict disease-related outcomes

ELIGIBILITY:
Inclusion criteria:

* Genetically confirmed FSHD1 or clinical diagnosis of FSHD with characteristic findings on exam and an affected parent or offspring (40)
* Age 18-75 years
* Symptomatic limb weakness
* Patient able to walk alone or with a walking aid.
* Patient affiliated to the social security system
* Patient giving written consent after written and oral information.
* If taking over the counter supplements willing to remain consistent with supplement regimen throughout the course of the study

Non inclusion criteria:

* Patients with comorbidity not related to the disease that can modify the natural evolution of the disease or would interfere with safe testing in the opinion of the Investigator
* Regular use of available muscle anabolic/catabolic agents such as corticosteroids, oral testosterone or derivatives, or oral beta agonists
* Use of an experimental drug in an FSHD clinical trial within the past 30 days
* Pregnant or nursing women for women of childbearing age
* Patient protected by law, under guardianship or curator ship, or not able to participate in a clinical study according to the article L.1121-16 of the French Public Health Code

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the patients' adherence to the program, with the mobile application, over 12 months | up to 12 months
  The adherence to the program will be evaluated based on the number of times a patient has performed a task without a reminder from the medical team compare to the number of total tasks to perform.

SECONDARY OUTCOMES:
Evaluate the global technical feasibility of remote assessment, using digital clinical outcome measures (COMs), in ambulant FSHD1 patients, over 12 months, from health care providers' perspective | up to 12 months
  The technical feasibility, from the physician perspective will be evaluated using a feasibility questionnaire containing several items, such as quality of the videos, completeness of the questionnaires, data storage and data transmission. This questionnaire will be filled every 6 months by the physician. Each item will be evaluated using a 2-point Likert scale, with two options (yes and no). The percentage of questionnaires with a score of 4/4 will be calculated and the overall technical feasibility from the physician's perspective will be achieved if at least 50% of the questionnaires have received a score of 4/4.
Evaluate the global technical feasibility of remote assessment, using digital clinical outcome measures (COMs), in ambulant FSHD1 patients, over 12 months, from patients' perspective | up to 12 months
  The technical feasibility, from the patient's perspective will be evaluated using a feasibility questionnaire containing several items, such as visibility, ease to use, clarity, stability, satisfaction. Each item will be evaluated using a 10-point Likert scale ranging from 1 to 10. Each individual score will be added to obtain a total sum score for the questionnaire. We will then calculate the total mean of all questionnaires and consider that the overall technical feasibility from the patients' perspective has been achieved if the total mean is at least 6/10.

OTHER OUTCOMES:
Evaluate the reliability of remote assessment, using the 1-minute Sit To Stand test (1 MSTST), in ambulant FSHD1 patients, over 12 months | up to 12 months
  The 1-minute Sit To Stand test (1 MSTST) collected at home or at the hospital will be compared to evaluate the reliability of the remote assessment in ambulant FSHD1 patients. The 1-minute Sit To Stand test (1 MSTST) will be documented at each study visit at hospital (T0, T6, and T12 months). Within a week after the hospital visit, the same test (1-minute Sit To Stand test (1 MSTST)) will be documented at the patients' home. Once the videos are recorded, a healthcare provider from the medical team will evaluate the video using a questionnaire to assess the reliability of the assessment. This questionnaire contains several items suc as instructions, usefulness, robustness, validation.
Evaluate the reliability of remote assessment, using the 1-minute Overhead arm elevation test (1 OAE), in ambulant FSHD1 patients, over 12 months | up to 12 months
  The 1-minute Overhead arm elevation test (1 OAE) collected at home or at the hospital will be compared to evaluate the reliability of the remote assessment in ambulant FSHD1 patients. The 1-minute Overhead arm elevation test (1 OAE) will be documented at each study visit at hospital (T0, T6, and T12 months). Within a week after the hospital visit, the same test (1-minute Overhead arm elevation test (1 OAE)) will be documented at the patients' home. Once the videos are recorded, a healthcare provider from the medical team will evaluate the video using a questionnaire to assess the reliability of the assessment. This questionnaire contains several items suc as instructions, usefulness, robustness, validation.
Evaluate the reliability of remote assessment, using the Digital Functional Region (DFR) exercises (with or without weight), in ambulant FSHD1 patients, over 12 months | up to 12 months
  The Digital Functional Region (DFR) exercises (with or without weight) collected at home or at the hospital will be compared to evaluate the reliability of the remote assessment in ambulant FSHD1 patients. The Digital Functional Region (DFR) exercises (with or without weight) will be documented at each study visit at hospital (T0, T6, and T12 months). Within a week after the hospital visit, the same test (Digital Functional Region (DFR) exercises (with or without weight)) will be documented at the patients' home. Once the videos are recorded, a healthcare provider from the medical team will evaluate the video using a questionnaire to assess the reliability of the assessment. This questionnaire contains several items suc as instructions, usefulness, robustness, validation.
Compare the robustness of the Digital Functional Region (DFR) exercises (with or without weight) compared to commonly used Reachable Work Space (RWS) in this population | up to 12 months
  The robustness of the new proposed COMs (full body motion video) to other FSHD outcomes commonly used to follow disease evolution (i.e., Reachable Workspace with and without weights) will be evaluated over 12 months. The results of the DFR will be compared to the results of the RWS to ensure DFR reliability.
Collect real life data on fatigue using a visual and analog scale for fatigue | up to 12 months
  Fatigue felt will be assessed with a visual and analog scale for fatigue. The scale ranges from 0 (no fatigue) to 10 (maximum thinkable fatigue). This evaluation will be completed every day during one-week per month, during 12 months
Collect real life data on pain using a visual and analog scale for pain. | up to 12 months
  Pain felt will be assessed with a visual and analog scale for pain. The scale ranges from 0 (no pain) to 10 (maximum thinkable pain). This evaluation will be completed every day during one-week per month, during 12 months
Collect real life data on sleep using a visual and analog scale for Sleep | up to 12 months
  Sleep felt will be assessed with a visual and analog scale for Sleep. The scale ranges from 0 (no sleep) to 10 (maximum thinkable sleep). This evaluation will be completed every day during one-week per month, during 12 months
Collect real life data on physical activity | up to 12 months
  Physical activity will be assessed by a specific questionnaire, completed every day during one-week per month. This questionnaire assess if the patient has performed a physical activity during the day, the type and the length of the activity.
Collect real life data on physical activity, using the the Recent Physical Activity Questionnaire (RPAQ) | up to 12 months
  RPAQ is splitted in 3 parts: physical activity within and around the house, travel to and from work and your work activity and hobbies. This questionnaire assess:
  * physical activity level (inactive if score is less than 8.3 Metabolic Equivalent of Task (MET).h/week, moderate if score ranges from 8.3 to 16.7 MET.h/week or high physical activity if score is greater than 16.7 MET.h/week)
  * sedentary time (settled is score is greater than 7 hours per day or not settled if score is less than or equal to 7 hours per day).
  The questionnaire RPAQ will be completed every 2 months during 12 months.
Collect real life data on quality of life, using the Quality of Life in genetic Neuromuscular Disease (QoL-gNMD) | up to 12 months
  The Quality of Life in Genetic Neuromuscular Disease Questionnaire (QOL-gNMD) is splitted in 3 domains: "Impact of Physical Symptoms" (score from 0 to 19), "Self-perception" (score from 0 to 24) and "Activities and Social Participation" (score from 0 to 27). It will be completed every 6 months, during 12 months
Collect real life data on socio-economic burden of the disease, using the WHO Disability Assessment Schedule 2.0 (WHODAS2.0) | up to 12 months
  The WHO Disability Assessment Schedule 2.0 (WHODAS2.0) is splitted in 6 domains of functioning, including cognition, mobility, self-care, getting along, life activities and participation. For each items, a score will be assigned by the patient, between "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4). The total score ranges from 0 (no disability) to 100 (full disability). The WHODAS2.0 will be completed every 6 months during 12 months.
Collect real life data on fatigue using the Fatigue Severity Scale (FSS) | up to 12 months
  The Fatigue Severity Scale (FSS) is a unidimensional scale which focuses on the physical aspects of fatigue. It is a self-reported questionnaire developed to measure the impact of disabling fatigue on daily functioning. It covers several areas including physical, social, and cognitive effects. The FSS is a patient-reported outcome composed of 9-items with scores ranging from 1 = "strongly disagree" to 7 = "strongly agree". The questionnaire FSS will be completed every 2 months, during 12 months
Collect real life data on physical activity, using the Work Productivity and Activity Impairment Questionnaire (WPAI) | up to 12 months
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a self-reported instrument to measure impairments in both paid work and unpaid work. It measures absenteeism, presentism as well as the impairments in unpaid activity because of health problem during the past seven days. It is compose by 6 questions allowing to derive four main outcomes: 1) percent work time missed due to health for those who were currently employed; 2) percent impairment while working due to health for those who were currently employed and actually worked in the past seven days; 3) percent overall work impairment due to health or those who were currently employed; and 4) percent activity impairment due to health for all respondents. The questionnaire WPAI will be completed every 2 months during 12 months.
Collect real life data on socio-economic burden of the disease, using the Modified Patient's Global Impression of Change (mPGIC) | up to 12 months
  The Modified Patient's Global Impression of Change (mPGIC) is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. The scale ranges from 1 (Very much improved) to 7 (very much worse). The mPGIC will be completed every 6 months during 12 months.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Lille, Lille, Hauts-de-France
  - CHU de Nice, Nice, Provence-Alpes-Côte d'Azur Region
  - Institut de Myologie, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No